CLINICAL TRIAL: NCT04512664
Title: Principal Investigator
Brief Title: Different Cold Application Times on Ecchmosis, Edema and Pain After Rhinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Eda Tekin, Register nurse, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: beykent
Record Dates: First submitted 2019-11-25; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Rhinoplasty; Cryotherapy Effect; Nurse's Role

STUDY DESIGN:
Intervention Model Description: Prospective, 2-group, Single-blind, Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short term group (Active Comparator): cold treatment for 4 hours
  Interventions: Other: cold application
- long term group (Experimental): cold treatment for 48 hours
  Interventions: Other: cold application

INTERVENTIONS:
Other: cold application — cold application with gel pacs

SUMMARY:
The aim of this study is to investigate the effects of different cold application times with cold gel pads after rhinoplasty on eyelid edema, eye ecchymosis and pain. A total of 60 patients undergoing rhinoplasty were divided into two groups by simple randomization method. Cold application applied to short term group for 4 hours and to long term group for 48 hours. Cold application was applied around both eyes with cold gel pads for 20 minutes per hour. Pain was evaluated with the Visuel Analog Scale, ecchymosis with eyelid ecchymosis score, and edema with eye-edema score. Edema and ecchymosis were evaluated on the 1st and 4th hours and 2nd day. Pain conditions were evaluated before and after analgesics for 1, 4 hours and 2 times daily.

DETAILED DESCRIPTION:
The research was carried out between January 2015 and March 2017 in an education and research hospital with a capacity of 26 beds. The research was suspended between July 2015 and January 2016. Patients who underwent rhinoplasty / septorhinoplasty operation between January 2015 and March 2017 with open or closed technique were included in the study. The study included patients who were 18 years of age or older who underwent a rhinoplasty / septorhinoplasty operation voluntarily. Patients who had cold allergy, refused to participate, applied outside of the research protocol and required re-operation in the early postoperative period due to complications were excluded from the study. All patients were provided with training and brochures for preoperative, intraoperative and postoperative periods. The cold application was done with gel pads of the same size and weight (13 cm x 13 cm-approximately 100 g) for 20 minutes per hour. Cold application was performed by the researcher in both groups for the first 4 hours. The patients in the short-term cold application group were given cold application by the researcher for 4 hours and 20 minutes per hour and the cold application was terminated. In the long-term application group, the first 4 hours of cold application were done by the researcher. Cold application after 4 hours; jel pads was applied at home by the patient's relative in accordance with the training given on the cold application protocol.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* who underwent rhinoplasty / septorhinoplasty
* voluntarily participated in the study

Exclusion Criteria:

* Patients with cold allergy,
* refused to participate,
* performed outside the research protocol,
* required early re-operation due to postoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Echymosis around the eye as assessed using 4-point Eyelid ecchmosis scale: Postoperative 1st hour | Postoperative 1st hour
  Bruising around the eye
Echymosis around the eye as assessed using 4-point Eyelid ecchmosis scale: Postoperative 4th hour | Postoperative 4th hour
  Bruising around the eye
Echymosis around the eye as assessed using 4-point Eyelid ecchmosis scale: Postoperative 2nd day | Postoperative 2nd day
  Bruising around the eye

SECONDARY OUTCOMES:
Edema around the eye as assessed using 4-point Eyelid edema scale: Postoperative 1st hour | postoperative 1st hour
  eyelid swelling
Edema around the eye as assessed using 4-point Eyelid edema scale: Postoperative 4th hour | postoperative 4th hour
  eyelid swelling
Edema around the eye as assessed using 4-point Eyelid edema scale: Postoperative 2nd day | postoperative 2nd day
  eyelid swelling

OTHER OUTCOMES:
Surgical Site Pain as assesed using 100 point-VAS: postoperative 1st hour | postoperative 1st hour
  Surgical site pain
Surgical Site Pain as assesed using 100 point-VAS: postoperative 4th hour | postoperative 4th hour
  Surgical site pain
Surgical Site Pain as assesed using 100 point-VAS: postoperative 1st day morning before take the analgesic | postoperative 1st day morning before take the analgesic
  Surgical site pain
Surgical Site Pain as assesed using 100 point-VAS: postoperative 1st day morning after take the analgesic | postoperative 1st day morning, 45 minutes after take the analgesic
  Surgical site pain
Surgical Site Pain as assesed using 100 point-VAS: postoperative 1st day evening, before take the analgesic | postoperative 1st day evening, before take the analgesic
  Surgical site pain
Surgical Site Pain as assesed using 100 point-VAS: postoperative 1st day evening after take the analgesic | postoperative 1st day evening, 45 minutes after take the analgesic
  Surgical site pain
Surgical Site Pain as assesed using 100 point-VAS: postoperative 2nd day morning before take the analgesic | postoperative 2nd day morning before take the analgesic
  Surgical site pain
Surgical Site Pain as assesed using 100 point-VAS: postoperative 2nd day after before take the analgesic | postoperative 2nd day after 45 minutes before take the analgesic
  Surgical site pain

CONTACTS AND LOCATIONS:
Overall Officials: YASEMİN EDA TEKİN, PHD, Principal Investigator — FACULTY MEMBER